CLINICAL TRIAL: NCT03377673
Title: Right Ventricular Geometry, Function, Morphology and Pulmonary Arterial Stiffness and Size Evaluation by Cardiac Magnetic Resonance
Brief Title: Right Ventricular and Pulmonary Artery Evaluation by CMR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Egle Ereminiene, Clinical Professor, Lithuanian University of Health Sciences
Other Study IDs: no. BE-2-23
Record Dates: First submitted 2017-12-06; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CMR — CMR is performed using a 1,5T whole-body system (Siemens Aera, Siemens Medical Solutions; Erlangen, Germany)

SUMMARY:
Pulmonary hypertension results in right ventricle dysfunction. Cardiac magnetic resonance derived RV ejection fraction is a prognostic value in this condition.

Right ventricular geometry, function, morphology as well as pulmonary arterial stiffness and size may be evaluated by cardiac magnetic resonance imaging and could have great importance in evaluation of pulmonary hypertension prognosis and outcomes.

DETAILED DESCRIPTION:
Pulmonary hypertension is defined as an increase in mean pulmonary artery pressure > 25 mmHg evaluated by right heart catheterisation. Over time increased pulmonary artery pressure eventually causes vascular remodelling and right ventricular dysfunction. The right and left ventricles interact sharing a common pericardial sac and interventricular septum. Frequently right ventricle dysfunction reflects clinical PH worsening.

The aim of this study was to assess the geometry, function and morphology of right ventricle and also pulmonary artery diameter and stiffness in pulmonary hypertension patients by cardiovascular magnetic resonance.

Patients are recruited from the Hospital of Lithuanian University of Health Sciences Kaunas clinics Pulmonary hypertension center.

Study inclusion criteria:

1. Patient with diagnosed pulmonary hypertension
2. RHC, 6MWT, echocardiography, NT-pro BNP, CMR performed in one month period.
3. Patients who signed study informed consent form.

Study exclusion criteria:

1. Coronary and valvular heart disease
2. Atrial fibrillation
3. Expressed shortness of breath
4. Claustrophobia.

Suspected number of participants - 100.

Data Analysis Statistical analyses will be performed using SPSS 22.0 package (SPSS, Chicago, IL, USA). Continuous variables will be expressed as mean +/- standard deviation, skewed variables as median (interquartile range). Chi square test will be used for qualitative parameters. For continuous variables, differences between two groups will be compared using non-parametric Mann-Whitney U test. Relation between variables will be assessed using Spearman correlation coefficient. Univariate analysis of predictors for survival will be used. In order to assess minimally false negative and minimally false positive results with greatest accuracy, the method of ROC (Receiver Operating Characteristics) curve will be used. The optimal values will be separated out the different groups (survival/non-survival) with the highest accuracy (minimal false negative and false positive). Survival curves will be established by the Kaplan-Meier estimation method. Cox regression analysis will be used to identify independent predictor of outcomes. Two-tailed probability values at p<0,05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with diagnosed pulmonary hypertension
2. RHC, 6MWT, echocardiography, NT-pro BNP, CMR performed in one month period.
3. Patients who signed study informed consent form.

Exclusion Criteria:

1. Coronary and valvular heart disease
2. Atrial fibrillation
3. Expressed shortness of breath
4. Claustrophobia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Precapillary pulmonary hypertesnion patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Right ventricle function and morphological changes in pulmonary hypertension patients during follow up | 2 years
  Right ventricle function will be evaluated by CMR at base line and during follow up to find significant values for disease progression and prognosis
Right ventricle function and morphological changes in pulmonary hypertension patients during follow up | 2 years
  Pulmonary artery will be evaluated by CMR at base line and during follow up to find significant values for disease progression and prognosis
Left ventricle function and mechanical changes in pulmonary hypertension patients during follow up | 2 years
  Left ventricle function and mechanical changes will be evaluated by CMR and FT at base line and during follow up to find significant values for disease progression and prognosis
Right ventricle mechanical changes in pulmonary hypertension patients during follow up | 2 years
  Right ventricle function and mechanical changes will be evaluated by FT at base line and during follow up to find significant values for disease progression and prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Lina Padervinskiene, PhD, Study Director — LSMU
Locations (1):
- LSMU, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided